CLINICAL TRIAL: NCT03344939
Title: Impact of Parent's Presence in Neonatology
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: NEONATLANUIT
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2017-11

CONDITIONS: Newborn; Vitality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Every year 75000 new-born babies are hospitalized in neonatology yard in France with about 60000 born prematurely.

Studies showed that parents presence is good for the baby development , decrease the stress due to hospitalization.It's also efficient for the attachment between the baby and parents.

Although the team try to settle a good atmosphere to establish this link and let parents take their position,it seems that the time taken to stay with the baby is less moreover the night.

The aim of the study is to evaluate the time of presence to find tools to increase this time in the neonatotology yard

ELIGIBILITY:
Inclusion Criteria:

* every newborn baby hospitalized in neonatology yard

Exclusion Criteria:

* no french speaking parents
* duration of hospitalization less than 1 week.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: every newborn baby hospitalized in neonatology yard
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
number of hours spent with the newborn baby the night. | Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France